CLINICAL TRIAL: NCT04192422
Title: Glucose Control and Metabolic Adaptation in Offspring of Women With Gestational Diabetes Recruited to the DiGest Study
Brief Title: DiGESTnewborn Study
Acronym: DiGESTnewborn
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kathryn Beardsall, Principle Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: DiGestnewborn v2.0 24.10.2019
Record Dates: First submitted 2019-11-29; First posted 2019-12-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: GDM; Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention — This is a cohort study no intervention

SUMMARY:
We wish to study the effect of a mothers sugar (glucose) control during pregnancy on her baby's sugar control after birth.

ELIGIBILITY:
Inclusion Criteria:

* mothers and their babies who have been enrolled in DiGest Trial and who have provided informed consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers and their babies who have been enrolled in DiGest Trial a trial of dietary intervention in women with gestational diabetes
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal sensor glucose time in target | From sensor insertion for up to the first 7 days of life
  Time sensor glucose levels in target in the first week of life

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrookes Hospital, Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No